CLINICAL TRIAL: NCT05747573
Title: An Open-label, Randomized, Three-period, Crossover Study to Compare the Pharmacokinetics of GB1211 Upon Dosing a Capsule Under Fasting Condition and a Tablet Under Fasting and Fed Conditions in Healthy Volunteers
Brief Title: A Study to Compare Pharmacokinetics of GB1211
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galecto Biotech AB (Industry)
Collaborators: QPS Holdings LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GALBA-1; GB1211-CPH-005 (Other: Galecto Biotech)
Record Dates: First submitted 2023-01-26; First posted 2023-02-28 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-02

CONDITIONS: Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A 100mg GB1211 tablet, fasted (Active Comparator): Single dose of 100 mg GB1211 as a tablet (100 mg strength) under fasted conditions (n=4 per period)
  Interventions: Drug: GB1211
- B 100 mg GB1211 capsules, fasted (Active Comparator): Single dose of 100 mg GB1211 as two capsules (50 mg strength) under fasted conditions (n=4 per period)
  Interventions: Drug: GB1211
- C 100 mg GB1211 tablet, fed (Active Comparator): Single dose of 100 mg GB1211 as a tablet (100 mg strength) under fed conditions (n=4 per period)
  Interventions: Drug: GB1211

INTERVENTIONS:
Drug: GB1211 — Hard tablet or capsules for oral use

SUMMARY:
This study is an open label, Randomized, Three-period, Crossover Study to Compare the Pharmacokinetics of GB1211 upon Dosing a Capsule under Fasting Condition and a Tablet under Fasting and Fed Conditions in Healthy Volunteers

DETAILED DESCRIPTION:
This is relative bioavailability and food effect study to enable further clinical development of a tablet formulation of GB1211.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide written informed consent prior to any Screening procedures being performed.
2. Male and female subjects 18-55 years of age (inclusive) on the day of signing the informed consent.
3. Subjects deemed in good physical health by the Investigator, as determined by no clinically significant findings from medical history, laboratory safety tests (serology, hematology, biochemistry and urinalysis), physical examination, vital signs, and electrocardiogram (ECG).
4. Women of child-bearing potential (WOCP) must agree not to attempt to become pregnant or donate ova, and to use a highly effective form of hormonal or non-hormonal birth control during the study and for 180 days after the last study drug administration, including:

   * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

     * oral
     * intravaginal
     * transdermal
   * progestogen-only hormonal contraception associated with inhibition of ovulation:

     * oral
     * injectable
     * implantable
   * intrauterine device (IUD)
   * intrauterine hormone-releasing system (IUS)
   * bilateral tubal occlusion
   * vasectomized partner
   * sexual abstinence
5. Postmenopausal women must have had ≥12 months of spontaneous amenorrhea (with documented follicle-stimulating hormone (FSH) ≥30 mIU/mL). Surgically sterile women are defined as those who have had a hysterectomy, bilateral ovariectomy, or bilateral tubal ligation. Women who are surgically sterile must provide documentation of the procedure.
6. Sexually active male subjects must use a barrier method of contraception (condom) and refrain from sperm donation during the study and for at least 90 days after the last study drug administration if their female sexual partner is of childbearing potential. Acceptable methods of birth control for female partners of male subjects are: hormonal contraceptives (oral contraceptives, implant or injection), intrauterine device (placed at least 1 month before the start of the study). Surgical sterilization of male patients can be accepted as a form of birth control if the sterilization procedure took place at least 6 months prior to the start of the study.
7. Adequate venous access for blood sampling.
8. Body mass index (BMI) between 18.0 to 32.0 kg/m2 (inclusive) at Screening.
9. Body temperature between 35.5-37.5 ºC (inclusive) at Screening and on Day -1 of Study Period 1.
10. Subjects agree to be available for the entire duration of the study and to be able to adhere to the study restrictions and examination schedule.
11. Able to swallow medication.
12. Subjects must be able to communicate well with the investigator and to comply with the requirements of the entire study.

Exclusion Criteria:

1. Contraindication or hypersensitivity to any drug or metabolites from similar class as study drug or to any excipients of the study drug formulation (including lactose).
2. Donation of 400 mL or more of blood or plasma within 8 weeks prior to first dosing.
3. Receipt of an investigational product within 90 days prior to the first dose of study drug.
4. History or presence of clinically significant ECG abnormalities or a family history or presence of prolonged QT-interval syndrome. Screening or Day -1 of Study Period 1 ECG: QTcF >450msec; PR >210 msec; QRS complex >119 msec, or other morphological changes other than repolarization, nonspecific S-T or T-wave changes.
5. Abnormal vital signs, after 5 minutes supine rest at Screening or on Day -1 of Study Period 1, defined as any of the following:

   1. Systolic blood pressure of < 90 or > 140 mmHg
   2. Diastolic blood pressure of < 45 or > 90 mmHg
   3. Pulse rate < 40 or > 100 bpm One (1) re-test may be performed at Screening and Day -1 of Study Period 1.
6. History of cardiac disease such as:

   1. Presence of clinically significant ventricular or atrial arrhythmia;
   2. History of clinically documented myocardial infarction;
   3. History of unstable angina pectoris;
   4. Other clinically significant cardiovascular disease (e.g., congestive heart failure).
7. Any positive result at Screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV), and on Day -1 for COVID-19.
8. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs. The investigator is to be guided by evidence of any of the following: history of major gastrointestinal surgery such as gastrectomy, gastroenterostomy, bowel resection or cholecystectomy. Subjects with a history of appendectomy are eligible to participate.
9. History of psychiatric illness within the past 2 years that may interfere with the ability to comply with the protocol requirements.
10. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in situ cervical cancer), treated or untreated, within 5 years, regardless of whether there is recurrence or metastases.
11. Smokers (use of tobacco or nicotine-containing products in the previous 3 months) and not willing to abstain from using tobacco or nicotine-containing products during the study. Positive cotinine test results at Screening or Day -1 are reason for exclusion. One (1) cotinine re-test may be performed at Screening and on Day -1 for otherwise eligible subjects who were recently exposed to passive smoke inhalation.
12. History of drug or alcohol abuse within 12 months prior to first dose and/or a positive urine drug screen/alcohol breath test at Screening or Day -1 of Study Period 1.
13. Use of any prescription or non-prescription medication including vaccination (excluding paracetamol, hormonal contraceptives), herbal medication, dietary supplements, or vitamins within 14 days prior to first dosing.
14. Administration of CYP3A4/5 inhibitors or inducers within 4 weeks prior to first dosing.
15. Administration of P-gp inhibitors or inducers within 4 weeks prior to first dosing.
16. Administration of medications that prolong the QT interval within 4 weeks prior to first dosing.
17. A positive pregnancy test at Screening or Day -1 of Study Period 1 or lactation.
18. Potentially unreliable or vulnerable subjects (e.g., person kept in detention) and those judged by the investigator to be unsuitable for the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
To measure the maximum plasma concentration of GB1211 (Cmax) | 5 weeks
  Timepoints for PK sampling
  Period 1: Day 1: pre-dose and at hrs 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24 (Day 2), 48 (Day 3), 72 (Day 4), and 96 (Day 5) post-dose.
  Period 2: Day 1: pre-dose and at 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24 (Day 2), 48 (Day 3), 72 (Day 4), and 96 (Day 5) post-dose.
  Period 3: Day 1: pre-dose and at 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24 (Day 2), 48 (Day 3), 72 (Day 4), and 96 (Day 5) post-dose.
To measure the time to reach Cmax GB1211 (Tmax) | 5 weeks
  Timepoints for PK sampling
  Period 1: Day 1: pre-dose and at hrs 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24 (Day 2), 48 (Day 3), 72 (Day 4), and 96 (Day 5) post-dose.
  Period 2: Day 1: pre-dose and at 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24 (Day 2), 48 (Day 3), 72 (Day 4), and 96 (Day 5) post-dose.
  Period 3: Day 1: pre-dose and at 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24 (Day 2), 48 (Day 3), 72 (Day 4), and 96 (Day 5) post-dose.
To measure the area under the plasma concentration-time curve of GB1211 (AUC) | 5 weeks
  Timepoints for PK sampling for
  Period 1: Day 1: pre-dose and at hrs 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24 (Day 2), 48 (Day 3), 72 (Day 4), and 96 (Day 5) post-dose.
  Period 2: Day 1: pre-dose and at 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24 (Day 2), 48 (Day 3), 72 (Day 4), and 96 (Day 5) post-dose.
  Period 3: Day 1: pre-dose and at 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24 (Day 2), 48 (Day 3), 72 (Day 4), and 96 (Day 5) post-dose.
To measure the amount of GB1211 excreted in urine (Ae) | 5 days
  Study Period 1: Pre-dose (single sample) and at [0 to 6 h], [6 to 12 h] (Day 1), [12 to 24 h] (Day 2), [24 to 48 h] (Day 3), [48 to 72 h] (Day 4), [72 to 96 h] (Day 5) post-dose.
To measure the fraction of GB1211 excreted in urine (Fe) | 5 days
  Study Period 1: Pre-dose (single sample) and at [0 to 6 h], [6 to 12 h] (Day 1), [12 to 24 h] (Day 2), [24 to 48 h] (Day 3), [48 to 72 h] (Day 4), [72 to 96 h] (Day 5) post-dose.

SECONDARY OUTCOMES:
To determine the number of participants with adverse events | 5 weeks
  Number of participants with adverse events graded as mild, moderate, or severe according to the study protocol.
  Number of participants with adverse events related and not related to the study drug.

OTHER OUTCOMES:
To determine the relative abundance of GB1211 metabolites in plasma and in urine | 5 weeks
  Plasma samples: Period 1: Day 1: pre-dose and at hrs 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24 (Day 2), 48 (Day 3), 72 (Day 4), and 96 (Day 5) post-dose.
  Period 2: Day 1: pre-dose and at 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24 (Day 2), 48 (Day 3), 72 (Day 4), and 96 (Day 5) post-dose.
  Period 3: Day 1: pre-dose and at 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24 (Day 2), 48 (Day 3), 72 (Day 4), and 96 (Day 5) post-dose.
  Urine samples: Study Period 1: Pre-dose (single sample) and at [0 to 6 h], [6 to 12 h] (Day 1), [12 to 24 h] (Day 2), [24 to 48 h] (Day 3), [48 to 72 h] (Day 4), [72 to 96 h] (Day 5) post-dose.

CONTACTS AND LOCATIONS:
Locations (1):
- QPS Netherlands BV, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aslanis V, Abd-Elaziz K, Slack RJ, Brinch A, Gravelle L, Morley W, Phung D, Herman K, Holyer I, Poulsen KK, Dogterom P, Tantawi S, Zetterberg FR, Jacoby B, Schambye H, Lindmark B. Relative bioavailability and food effect of the galectin-3 inhibitor selvigaltin (GB1211) administered as a tablet in healthy participants (GALBA-1). Cancer Chemother Pharmacol. 2024 Nov;94(5):707-720. doi: 10.1007/s00280-024-04710-3. Epub 2024 Aug 21. PMID 39167148